CLINICAL TRIAL: NCT05608928
Title: Ability of the Probiotic Vivomixx to Improve Environmental Enteropathy in Pregnant Women: a Proof of Concept Trial in Bangladesh, Pakistan, Senegal and Zambia
Acronym: EMP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tropical Gastroenterology & Nutrition Group (TROPGAN) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: NHRA000014/18/07/2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Environmental Enteropathy

STUDY DESIGN:
Intervention Model Description: Multi-site phase II randomised controlled trial
Who Masked: Participant, Investigator
Masking Description: Vivomixx and placebo drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vivomixx (Experimental): Vivomixx also known as VSL#3 is a commercial probiotic mixture consisting of eight probiotic lactic acid bacteria and Bifidobacteria including Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus casei, Lactobacillus delbrueckii subspecies bulgaricus, Streptococcus salivarius subspecies thermophiles, Bifidobacterium breve, Bifidobacterium longum, and Bifidobacterium infantis. VSL#3 contributes to balancing the gut and vaginal microbiota and is used as a food supplement for management of diseases like irritable bowel syndrome, ulcerative colitis or ileal pouch.
  Interventions: Dietary Supplement: VSL#3; Device: Capscan device; Combination Product: Placebo
- Capscan device (Experimental): The CapScan device is a short-term single-use class IIa ingestible medical device that collects fluids from the gastrointestinal ("GI") tract and is collected in the stool. GI samples are then extracted from the device and analyzed outside the body.
  Interventions: Dietary Supplement: VSL#3; Device: Capscan device; Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 — VSL#3 is a commercial probiotic mixture consisting of eight probiotic lactic acid bacteria and Bifidobacteria including Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus casei, Lactobacillus delbrueckii subspecies bulgaricus, Streptococcus salivarius subspecies thermophiles, Bifidobacterium breve, Bifidobacterium longum, and Bifidobacterium infantis. VSL#3 contributes to balancing the gut and vaginal microbiota and is used as a food supplement for management of diseases like irritable bowel syndrome, ulcerative colitis or ileal pouch.
  Other Names: Vivomixx
Device: Capscan device — The CapScan device is a short-term single-use class IIa ingestible medical device that collects fluids from the gastrointestinal ("GI") tract and is collected in the stool. GI samples are then extracted from the device and analyzed outside the body.
  Other Names: capstan
Combination Product: Placebo — microcrystalline cellulose

SUMMARY:
This trial will determine if a well-established probiotic, Vivomixx, can modulate the maternal microbiota and ameliorate the maternal environmental enteropathy which compromises growth in the first 1000 days. The probiotic Vivomixx has been used in many thousands of people including pregnant women, both within and outside a research context. This trial is the first in a proposed series of proof-of-concept intervention studies which are intended to provide data to enable a rational selection of interventions to be evaluated at scale in future large scale phase 2 trial in which birth outcomes and postnatal growth will be key endpoints.

DETAILED DESCRIPTION:
Stunting in young children refers to attenuated linear growth1. In the year 2020, 149.2 million children under the age of 5 years of age were stunted, accounting for 22% of stunting globally2. Stunting has short- and long-term consequences of increased morbidity and mortality3,4, impairment of neurocognitive development5 , impaired responses to oral vaccines6,7, and increased risk of non-communicable diseases. Stunting is partly driven by Environmental Enteric Dysfunction (EED), an enteropathic condition characterised by altered gut permeability, infiltration of immune cells and changes in villous architecture and cell differentiation8,9. EED may help explain why nutritional supplementation either during pregnancy or early childhood has minimal value in correcting childhood stunting10,11 Indeed, EED is believed to be responsible for 40% of childhood stunting12. Disruption in intestinal barrier function affects gut immune homeostasis, nutrient flows, and consequently dysbiosis in the gut microbiome. The gut microbiota consists of 100 trillion bacteria which interact with epithelial cells, the mucus layer and the mucosal immune system that balances tolerance and effector functions. Thus the gut microbiome has an important role in shaping the responsiveness of the gut immune system13. The mucus barrier and the normal gut microbiota limit enteropathogen colonisation. Influx of bacteria from the lumen to the systemic circulation represents microbial translocation and initiation of systemic of inflammatory process through recognition of pathogen-associated molecular patterns (PAMPs) by Pattern Recognition Receptors (PRRs) present on Antigen Presenting Cells (APCs). Three fundamental processes drive the epithelial damage which is so important in EED: infection, undernutrition, and immune dysfunction. Multiple clinical trials show that efforts to correct malnutrition through conventional therapies and improving hygiene and sanitation do not overcome growth deficits by more than about 10%10,11. There is increasing interest in the use of probiotics which may allow pathogen decolonization, improve barrier function and restore overall gut homeostasis. Such therapies are at early stage of trials but may have potential in addressing the global burden of EED, by improving barrier function and gut pathophysiology.

Colonization of gut by enteropathogens is common in children with EED. These include ETEC, Campylobacter, Shigella and Salmonella species. Consistent data from Bangladesh and Zambia show that children with refractory stunting carry over four pathogens on average, whilst controls carry less than two14,15. There is also clear evidence of altered composition of the microbiota in children with EED16,17,18.

Probiotics may serve to overcome the problem of EED through all mechanisms of pathogenicity, by providing additional bacteria that may help in intestinal decolonization of pathogenic microorganisms (changing the microbiological niche), promoting epithelial healing, improving nutrient absorption, and restoration of an appropriate immune balance between tolerance and responsiveness.

To date the focus of research on childhood stunting has been on the young child. It is increasingly appreciated, however, that stunting often begins in utero and the focus has shifted to women's health and pregnancy. For example, the Lancet 2021 Series on maternal and child undernutrition states that "Investments to reduce undernutrition in women are important not only for women's own health but also for the health and nutrition of their children"19. Results from rural Bangladesh reveal poor gestational weight gain that ultimately leads to intrauterine growth restriction, low birth weight and ultimately stunting and wasting20,21. Furthermore, another study recently completed in slum settlements of Dhaka, Bangladesh demonstrated a high prevalence of EED among undernourished women. Intestinal histopathology was abnormal in more than 80% of women22. We postulate that growth retardation in utero is a consequence of EED in the mother during pregnancy and lactation. This leads to systemic inflammation, which leads to disadvantageous partitioning of nutrients, and reduced nutrient availability.

This trial will explore the conceptual framework that a well known probiotic, that can improve the composition of the gut microbiota, can also reduce biomarkers of intestinal inflammation and gut health. This will restore healthy microbial signalling to the host epithelium, ameliorate barrier function through secretion of mucus and antimicrobial factors, and improve nutrient availability.

ELIGIBILITY:
Inclusion Criteria:

Women over the age of 18 years in the second trimester of pregnancy, living in defined geographical areas of Bangladesh, Pakistan, Senegal and Zambia, where it can be assumed that environmental enteropathy is universal.

Exclusion Criteria

Potential participants will not be enrolled if they:

* have had diarrhoea, defined as the passage of three or more loose stools per 24 hours, in the preceding 14 days;
* have taken antibiotics or probiotics in the preceding 14 days;
* have taken non-steroidal anti-inflammatory drugs in the preceding 14 days;
* have haemoglobin concentration <8g/dl;
* have any illness which in the opinion of the investigator will complicate assessment of safety or efficacy;
* have any gastrointestinal contraindication to ingestion of a capsule (known or suspected gastrointestinal obstruction, stricture, fistula, gastroparesis, or any swallowing disorder);
* have a plan to leave the study area within the follow-up period;

but may be enrolled if/when these disqualifiers have expired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage change (mean, unweighted) in a multiple panel of biomarkers between baseline and last sample collected after 56 days of treatment, compared to control group. | 2 months
  Plasma CRP by ELISA Plasma AGP by ELISA Plasma sCD14 by ELISA Plasma LBP by ELISA Plasma iFABP by ELISA Plasma CD163 by ELISA Faecal MPO by ELISA Faecal neopterin by ELISA Faecal calprotectin by ELISA Faecal lipocalin by ELISA

SECONDARY OUTCOMES:
Reduction in colonisation | 2 Months
  Stool qPCR for Salmonella, Shigella, Campylobacter, ETEC, EPEC, EAEC, rotavirus, norovirus, Giardia and Cryptosporidium
Change in microbiome | 2 months
  Whole genome shotgun metagenomics sequencing (MetaPhlAn) in faecal and CAPSCAN samples
Reduction in LR ratio in Vivomixx compared to placebo groups | 2 months
  LR ratio in 3 hour/120 min urine collections following dose of 5g lactulose and 1g rhamnose
Change in metabolome | 2 months
  Untargeted urine and plasma (and fecal) metabolome before and after intervention
Weight gain velocity in the 2nd trimester of pregnancy | weekly for 56 days
  Rate of weight gain (kg/week)
Measurements of variability, including standard deviations and kappa values | 2 months
  Preliminary work across all sites using identical kits and harmonised SOPs

OTHER OUTCOMES:
Tertiary outcome:Recovery of useful data from CapScan | 2 months
  Completion of whole gut microbiome profiles

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kelly, Dr, Principal Investigator — Tropical Gastroenterology & Nutrition Group (TROPGAN); Yakhya Dieye, Dr, Principal Investigator — Institut Pasteur de Dakar; Fyezah Jehan, Dr, Principal Investigator — Aga Khan University; Asad Ali, Dr, Principal Investigator — Aga Khan University; Tahmeed Ahmed, Dr, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (4):
- Icddr,B, Dhaka, Bangladesh
- Aga Khan University, icddr,b, Karachi, Sindh, Pakistan
- Institut pasteur de dakar, Dakar, Senegal
- TROPGAN, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Olofin I, McDonald CM, Ezzati M, Flaxman S, Black RE, Fawzi WW, Caulfield LE, Danaei G; Nutrition Impact Model Study (anthropometry cohort pooling). Associations of suboptimal growth with all-cause and cause-specific mortality in children under five years: a pooled analysis of ten prospective studies. PLoS One. 2013 May 29;8(5):e64636. doi: 10.1371/journal.pone.0064636. Print 2013. PMID 23734210
- [Background] Prendergast AJ, Humphrey JH. The stunting syndrome in developing countries. Paediatr Int Child Health. 2014 Nov;34(4):250-65. doi: 10.1179/2046905514Y.0000000158. Epub 2014 Oct 13. PMID 25310000
- [Result] de Onis M, Branca F. Childhood stunting: a global perspective. Matern Child Nutr. 2016 May;12 Suppl 1(Suppl 1):12-26. doi: 10.1111/mcn.12231. PMID 27187907